CLINICAL TRIAL: NCT04366921
Title: European/Euro-ELSO Survey on Adult and Neonatal/ Pediatric COVID Patients in ECMO
Brief Title: European/Euro-ELSO Survey on Adult and Neonatal/ Pediatric COVID-19 Patients in ECMO
Acronym: EuroECMO-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: European chapter of the Extracorporeal Life Support Organization (Unknown); Erasmus Medical Center (Other); Leiden University Medical Center (Other); UMC Utrecht (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Papa Giovanni XXIII Hospital (Other); Niguarda Hospital (Other); Ospedale San Donato (Other); Ospedale S. Giovanni Bosco (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Ospedale dell'Angelo, Venezia-Mestre (Other); University Hospital, Udine, Italy (Other); San Gerardo Hospital (Other); Ospedali Riuniti Ancona (Other); San Camillo Hospital, Rome (Other); San Giorgio Clinic (Unknown); GVM Care & Research (Unknown); San Raffaele University Hospital, Italy (Other); Ospedale San Bortolo di Vicenza (Other); Klinik Hirslanden, Zurich (Other); University of Zurich (Other); Cardiocentro Ticino (Other); Vilnius University Hospital Santaros Klinikos (Other); University Düsseldorf (Other); Klinikum Nürnberg (Other); Hannover Medical School (Other); Heart Center Leipzig - University Hospital (Other); University Hospital Regensburg (Other); University Hospital, Essen (Other); German Heart Center (Other); University Hospital, Aachen (Other); University Heart Center Freiburg - Bad Krozingen (Other); Klinikum Kassel (Other); General University Hospital, Prague (Other); Universitaire Ziekenhuizen KU Leuven (Other); Onze Lieve Vrouwziekenhuis Aalst (Other); Erasme University Hospital (Other); University Hospital, Antwerp (Other); Hôpital Civil Marie Curie de Charleroi (Unknown); University Hospital, Ghent (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Hospital Vall d'Hebron (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Miguel Servet (Other); Henri Mondor University Hospital (Other); Hospices Civils de Lyon (Other); Pitié-Salpêtrière Hospital (Other); Rennes University Hospital (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Karolinska University Hospital (Other); Hospital Sao Joao (Other); Medical University of Warsaw (Other); Universitätskliniken Innsbruck (Unknown); Medical University of Vienna (Other); University Hospital, Alexandroupolis (Other); Novosibirsk City Hospital #2 (Other); City Clinical Hospital No. 67, Moscow, Russia (Other Government); City Hospital No 40, Saint Petersburg, Russia (Other); Krasnodar Regional Hospital no 1 (Unknown); Kemerovo Regional Clinical Cardiological Center named after academician L.S. Barbarash (Unknown); City Hospital No 41, Ekaterinburg, Russia (Other); G. Pasquinucci Heart Hospital, Massa (Other); Charles University, Czech Republic (Other); University Hospital, Bordeaux (Other); Bambino Gesù Hospital and Research Institute (Other); Policlinico Hospital Milan (Unknown); Gaslini Children's Hospital (Other); Children's Medical Hospital, University of Essen, Essen, Germany (Other); University Hospital, Geneva (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Paediatric Intensive Care Glasgow (Unknown); Paris South University Hospitals (Unknown); University of Groningen (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Hospital Sant Joan de Deu (Other); Heim Pal Children's Hospital (Other); University Hospital, Montpellier (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Lund University Hospital (Other); Landesklinikum Sankt Polten (Other); Chelyabinsk Regional Clinical Hospital (Other Government); ECMO Centers Israel (Unknown); Copenhagen University Hospital at Herlev (Other); Ospedale M. Bufalini Cesena (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); Mauriziano Umberto I Hospital (Other); University of Bern (Other); University Hospital, Basel, Switzerland (Other); University of Lausanne Hospitals (Other); University Hospital Tuebingen (Other); Universitätsklinikum Köln (Other); Chirec (Other); Universitair Ziekenhuis Brussel (Other); Centre Hospitalier Universitaire de Liege (Other); La Louvière Hopital (Unknown); Leicester Royal Infirmary NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2020-1343
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: COVID; SARS-CoV-2; ARDS, Human; Refractory Hypoxemia; Cardiogenic Shock; Septic Shock; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia; Shock, Cardiogenic; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the last 10 years, severe acute respiratory infection (SARI) was responsible of multiple outbreaks putting a strain on the public health worldwide. Indeed, SARI had a relevant role in the development of pandemic and epidemic with terrible consequences such as the 2009 H1N1 pandemic which led to more than 200.000 respiratory deaths globally.

In late December 2019, in Wuhan, Hubei, China, a new respiratory syndrome emerged with clinical signs of viral pneumonia and person-to-person transmission. Tests showed the appearance of a novel coronavirus, namely the 2019 novel coronavirus (COVID-19). Two other strains, the severe acute respiratory syndrome coronavirus (SARS-CoV) and Middle East respiratory syndrome coronavirus (MERS-CoV) have caused severe respiratory illnesses, sometimes fatal. In particular, the mortality rate associated with SARS-CoV and MERS-CoV, was of 10% and 37% respectively.

Even though COVID-19 appeared from the first time in China, quickly it spread worldwide and cases have been described in other countries such as Thailand, Japan, South Korea, Germany, Italy, France, Iran, USA and many other countries. An early paper reported 41 patients with laboratory-confirmed COVID-19 infection in Wuhan. The median age of the patients was 49 years and mostly men (73%). Among those, 32% were admitted to the ICU because of the severe hypoxemia. The most associated comorbidities were diabetes (20%), hypertension (15%), and cardiovascular diseases (15%). On admission, 98% of the patients had bilateral multiple lobular and sub-segmental areas of consolidation. Importantly, acute respiratory distress syndrome (ARDS) developed in 29% of the patients, while acute cardiac injury in 12%, and secondary infection in 10%. Invasive mechanical ventilation was required in 10% of those patients, and two of these patients (5%) had refractory hypoxemia and received extracorporeal membrane oxygenation (ECMO). In a later retrospective report by Wang and collaborators, clinical characteristics of 138 patients with COVID-19 infection were described. ICU admission was required in 26.1% of the patients for acute respiratory distress syndrome (61.1%), arrhythmia (44.4%), and shock (30.6%). ECMO support was needed in 11% of the patients admitted to the ICU. During the period of follow-up, overall mortality was 4.3%.

The use of ECMO in COVID-19 infection is increasing due to the high transmission rate of the infection and the respiratory-related mortality.

Therefore, the investigators believe that ECMO in case of severe interstitial pneumonia caused by COVID could represent a valid solution in order to avoid lung injuries related to prolonged treatment with non-invasive and invasive mechanical ventilation. In addition, ECMO could have a role for the systemic complications such as septic and cardiogenic shock as well myocarditis scenarios. Potential clinical effects and outcomes of the ECMO support in the novel coronavirus pandemic will be recorded and analyzed in our project.

The researchers hypothesize that a significant percentage of patients with COVID-19 infection will require the utilize of ECMO for refactory hypoxemia, cardiogenic shock or septic shock. This study seeks to prove this hypothesis by conducting an observational retrospective/prospective study of patients in the ICU who underwent ECMO support and describe clinical features, severity of pulmonary dysfunction and risk factors of COVID-patients who need ECMO support, the incidence of ECMO use, ECMO technical characteristics, duration of ECMO, complications and outcomes of COVID-patients requiring ECMO support.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed COVID-19 infection by real-time PCR (polymerase chain reaction)
* ECMO for treatment severe lung disease COVID-19 related

Exclusion Criteria:

* Patients treated with ECMO for other concomitant causes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with confirmed COVID-19 infection who require ECMO support
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Age | at baseline
  age in years
Gender | at baseline
  male/female
Weight | at baseline
  in kilograms
Height | at baseline
  in meters
BMI | at baseline
  weight and height combined to calculate BMI in kg/m^2
Pre-existing pulmonary disease y/n | at baseline
  Asthma y/n, cystic fibrosis y/n, chronic obstructive pulmonary disease y/n, pulmonary hypertension y/n, pulmonary fibrosis y/n, chronic restrictive lung disease y/n
Main co-morbidities y/n | at baseline
  diabetes mellitus y/n, chronic renal failure y/n, ischemic heart disease y/n, heart failure y/n, chronic liver failure y/n, neurological impairment y/n
Date of signs of COVID-19 infection | at baseline or date of occurence
  in dd-mm-yyyy or mm-dd-yyyy
Date of positive swab | at baseline or date of occurence
  in dd-mm-yyyy or mm-dd-yyyy
Pre-ECMO length of hospital stay | at or during ECMO-implant
  in days
Pre-ECMO length of ICU stay | at or during ECMO-implant
  in days
Pre-ECMO length of mechanical ventilation days | at or during ECMO-implant
  in days
Use of antibiotics | up to 6 months
  y/n, what kind
Use of anti-viral treatment | up to 6 months
  y/n, what kind
Use of second line treatment | up to 6 months
  y/n, what kind (eg prone-position, recruitment manoeuvers, neuromuscular blockade etc)
Indications for ECMO-implant | at ECMO-implant
  respiratory or cardiac
Type of ECMO-implant | at ECMO-implant
  veno-venous, veno-arterial or veno-venoarterial
Type of access | at ECMO-implant
  peripheral or central
Date of ECMO implant | at ECMO-implant
  in dd-mm-yyyy or mm-dd-yyyy
ECMO blood flow rate | from day of ECMO-implant for every 24 hours until date of weaning or death, up to 6 months
  l/min
ECMO gas flow rate | from day of ECMO-implant for every 24 hours until date of weaning or death, up to 6 months
  l/min
ECMO configuration change | up to 6 months
  y/n
Date of ECMO configuration change | up to 6 months
  in dd-mm-yyyy or mm-dd-yyyy
New ECMO configuration | up to 6 months
  veno-venous, veno-arterial, veno-venoarterial, other
Indications for ECMO configuration change | up to 6 months
  right ventricular failure, left ventricular failure, refractory hypoxemia
Ventilator setting on ECMO | from day of ECMO-implant for every 24 hours until date of weaning or death, up to 6 months
  settings of ventilator
Anticoagulation during ECMO | from day of ECMO-implant for every 24 hours until date of weaning or death, up to 6 months
  heparin, bivalirudin, nothing
Frequency of ECMO circuit change | up to 6 months
  amount of ECMO circuit changes (1, 2, 3 etc.)
ECMO complications | up to 6 months
  Hemorrhagic, infection, other complications
ECMO Weaning | from day of ECMO-implant for every 24 hours until date of weaning or death, up to 6 months
  y/n
ICU discharge | from day of ICU-admission for every 24 hours until date of discharge or death, up to 6 months
  y/n, date
Main cause of death | 6 months
Type of discharge | up to 6 months
  Ward, another ICU, rehabilitation center, home
Alive/deceased | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorusso, Prof. Dr., Principal Investigator — Maastricht University Hospital
Locations (97):
- Austria (3):
  - Universitätskliniken Innsbruck, Innsbruck
  - Landesklinikum Sankt Polten, Sankt Pölten
  - Medical University of Vienna, Vienna
- Belgium (11):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - University Hospital, Antwerp, Antwerp
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - Chirec, Brussels
  - Erasme University Hospital, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Hôpital Civil Marie Curie de Charleroi, Charleroi
  - University Hospital, Ghent, Ghent
  - La Louvière Hopital, La Louvière
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHU de Liege, Liège
- Czechia (2):
  - Charles University, Czech Republic, Prague
  - General University Hospital, Prague, Prague
- Copenhagen University Hospital at Herlev, Copenhagen, Denmark
- France (7):
  - University Hospital, Bordeaux, Bourdeaux
  - Hospices Civils de Lyon, Lyon
  - University Hospital, Montpellier, Montpellier
  - Henri Mondor University Hospital, Paris
  - Paris South University Hospitals, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Rennes University Hospital, Rennes
- Germany (13):
  - University Hospital, Aachen, Aachen
  - German Heart Center, Berlin
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Children's Medical Hospital, University of Essen, Essen, Germany, Essen
  - University Hospital, Essen, Essen
  - University Heart Center Freiburg - Bad Krozingen, Freiburg im Breisgau
  - Hannover Medical School, Hanover
  - Klinikum Kassel, Kassel
  - Heart Center Leipzig - University Hospital, Leipzig
  - Klinikum Nürnberg, Nuremberg
  - University Hospital Regensburg, Regensburg
  - University Hospital Tuebingen, Tübingen
- University Hospital, Alexandroupolis, Alexandroupoli, Greece
- Heim Pal Children's Hospital, Budapest, Hungary
- ECMO Centers Israel, Jerusalem, Israel
- Italy (23):
  - San Giorgio Clinic, Alessandria
  - Ospedali Riuniti Ancona, Ancona
  - Papa Giovanni XXIII Hospital, Bergamo
  - St. Orsola Hospital, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale Maurizio Bufalini, Cesena
  - Gaslini Children's Hospital, Genoa
  - G. Pasquinucci Heart Hospital, Massa, Massa
  - Niguarda Hospital, Milan
  - Ospedale San Donato, Milan
  - San Raffaele University Hospital, Italy, Milan
  - Policlinico Hospital Milan, Milan
  - San Gerardo Hospital, Monza
  - IRCCS Policlinico S. Matteo, Pavia
  - GVM Care & Research, Puglia
  - Bambino Gesù Hospital and Research Institute, Roma
  - San Camillo Hospital, Rome, Roma
  - A.O.U. Città della Salute e della Scienza - Molinette Hospital, Turin
  - Mauriziano Umberto I Hospital, Turin
  - Ospedale S. Giovanni Bosco, Turin
  - University Hospital, Udine, Italy, Udine
  - Ospedale dell'Angelo, Venezia-Mestre, Venice
  - Ospedale San Bortolo di Vicenza, Vicenza
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Netherlands (5):
  - University of Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht, Utrecht
- Medical University of Warsaw, Warsaw, Poland
- Hospital Sao Joao, Porto, Portugal
- Russia (7):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Kemerovo Regional Clinical Cardiological Center named after academician L.S. Barbarash, Kemerovo
  - Krasnodar Regional Hospital no 1, Krasnodar
  - City Clinical Hospital No. 67, Moscow, Russia, Moscow
  - Novosibirsk City Hospital #2, Novosibirsk
  - City Hospital No 40, Saint Petersburg, Russia, Saint Petersburg
  - City Hospital No 41, Ekaterinburg, Russia, Yekaterinburg
- Spain (4):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Miguel Servet, Zaragoza
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
- Switzerland (7):
  - University Hospital, Basel, Switzerland, Basel
  - University of Bern, Bern
  - University Hospital, Geneva, Geneva
  - University of Lausanne Hospitals, Lausanne
  - Cardiocentro Ticino, Lugano
  - Klinik Hirslanden, Zurich, Zurich
  - University of Zurich, Zurich
- United Kingdom (6):
  - Royal Brompton & Harefield NHS Foundation Trust, Brompton
  - Paediatric Intensive Care Glasgow, Glasgow
  - Leicester Children's Hospital, Leicester
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolotin S, Pebody R, White PJ, McMenamin J, Perera L, Nguyen-Van-Tam JS, Barlow T, Watson JM; UK Severe Influenza Surveillance System (USISS) Steering Group. A new sentinel surveillance system for severe influenza in England shows a shift in age distribution of hospitalised cases in the post-pandemic period. PLoS One. 2012;7(1):e30279. doi: 10.1371/journal.pone.0030279. Epub 2012 Jan 23. PMID 22291929
- [Background] Dawood FS, Iuliano AD, Reed C, Meltzer MI, Shay DK, Cheng PY, Bandaranayake D, Breiman RF, Brooks WA, Buchy P, Feikin DR, Fowler KB, Gordon A, Hien NT, Horby P, Huang QS, Katz MA, Krishnan A, Lal R, Montgomery JM, Molbak K, Pebody R, Presanis AM, Razuri H, Steens A, Tinoco YO, Wallinga J, Yu H, Vong S, Bresee J, Widdowson MA. Estimated global mortality associated with the first 12 months of 2009 pandemic influenza A H1N1 virus circulation: a modelling study. Lancet Infect Dis. 2012 Sep;12(9):687-95. doi: 10.1016/S1473-3099(12)70121-4. Epub 2012 Jun 26. PMID 22738893
- [Background] Simonsen L, Spreeuwenberg P, Lustig R, Taylor RJ, Fleming DM, Kroneman M, Van Kerkhove MD, Mounts AW, Paget WJ; GLaMOR Collaborating Teams. Global mortality estimates for the 2009 Influenza Pandemic from the GLaMOR project: a modeling study. PLoS Med. 2013 Nov;10(11):e1001558. doi: 10.1371/journal.pmed.1001558. Epub 2013 Nov 26. PMID 24302890
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Drosten C, Gunther S, Preiser W, van der Werf S, Brodt HR, Becker S, Rabenau H, Panning M, Kolesnikova L, Fouchier RA, Berger A, Burguiere AM, Cinatl J, Eickmann M, Escriou N, Grywna K, Kramme S, Manuguerra JC, Muller S, Rickerts V, Sturmer M, Vieth S, Klenk HD, Osterhaus AD, Schmitz H, Doerr HW. Identification of a novel coronavirus in patients with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1967-76. doi: 10.1056/NEJMoa030747. Epub 2003 Apr 10. PMID 12690091
- [Background] Ksiazek TG, Erdman D, Goldsmith CS, Zaki SR, Peret T, Emery S, Tong S, Urbani C, Comer JA, Lim W, Rollin PE, Dowell SF, Ling AE, Humphrey CD, Shieh WJ, Guarner J, Paddock CD, Rota P, Fields B, DeRisi J, Yang JY, Cox N, Hughes JM, LeDuc JW, Bellini WJ, Anderson LJ; SARS Working Group. A novel coronavirus associated with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1953-66. doi: 10.1056/NEJMoa030781. Epub 2003 Apr 10. PMID 12690092
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] de Groot RJ, Baker SC, Baric RS, Brown CS, Drosten C, Enjuanes L, Fouchier RA, Galiano M, Gorbalenya AE, Memish ZA, Perlman S, Poon LL, Snijder EJ, Stephens GM, Woo PC, Zaki AM, Zambon M, Ziebuhr J. Middle East respiratory syndrome coronavirus (MERS-CoV): announcement of the Coronavirus Study Group. J Virol. 2013 Jul;87(14):7790-2. doi: 10.1128/JVI.01244-13. Epub 2013 May 15. No abstract available. PMID 23678167
- [Background] Spina S, Marrazzo F, Migliari M, Stucchi R, Sforza A, Fumagalli R. The response of Milan's Emergency Medical System to the COVID-19 outbreak in Italy. Lancet. 2020 Mar 14;395(10227):e49-e50. doi: 10.1016/S0140-6736(20)30493-1. Epub 2020 Feb 28. No abstract available. PMID 32119824
- [Background] Ebrahim SH, Memish ZA. COVID-19: preparing for superspreader potential among Umrah pilgrims to Saudi Arabia. Lancet. 2020 Mar 14;395(10227):e48. doi: 10.1016/S0140-6736(20)30466-9. Epub 2020 Feb 27. No abstract available. PMID 32113506
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Derived] De Piero ME, Mariani S, van Bussel BCT, Jarczak D, Krenner N, de la Sota EP, Silva PE, Roemmer M, Kowalewski M, Carelli S, Broman LM, Vuylsteke A, Fortuna P, Alessandri F, Martucci G, Patel BV, Lotz G, Boeken U, Maier S, Filip B, Meyns B, Haenggi M, Puss S, Schellongowski P, Kirali K, Bolotin G, Barrett N, Riera J, Mueller T, Belohlavek J, Lorusso R; EuroECMO-COVID Study Group. In-hospital outcomes and 6-month follow-up results of patients supported with extracorporeal membrane oxygenation for COVID-19 from the second wave to the end of the pandemic (EuroECMO-COVID): a prospective, international, multicentre, observational study. Lancet Respir Med. 2025 Apr;13(4):307-317. doi: 10.1016/S2213-2600(24)00369-2. Epub 2025 Feb 23. PMID 40010369
- [Derived] Lorusso R, De Piero ME, Mariani S, Di Mauro M, Folliguet T, Taccone FS, Camporota L, Swol J, Wiedemann D, Belliato M, Broman LM, Vuylsteke A, Kassif Y, Scandroglio AM, Fanelli V, Gaudard P, Ledot S, Barker J, Boeken U, Maier S, Kersten A, Meyns B, Pozzi M, Pedersen FM, Schellongowski P, Kirali K, Barrett N, Riera J, Mueller T, Belohlavek J; EuroECMO-COVID Study Group. In-hospital and 6-month outcomes in patients with COVID-19 supported with extracorporeal membrane oxygenation (EuroECMO-COVID): a multicentre, prospective observational study. Lancet Respir Med. 2023 Feb;11(2):151-162. doi: 10.1016/S2213-2600(22)00403-9. Epub 2022 Nov 16. PMID 36402148